CLINICAL TRIAL: NCT06781242
Title: Genotype-phenotype Relationship Between Adult Cryptogenic Cholestasis and Mutations in Genes Responsible for Progressive Familial Intrahepatic Cholestasis
Brief Title: Genotype-phenotype Relationship Between Cryptogenic Cholestasis and Familial Intrahepatic Cholestasis
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: Ad-FIC; 3000468 (Other Grant/Funding Number: Albireo Pharma, Inc.)
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Cholestatic Liver Disease; Intrahepatic Cholestasis; Progressive Familial Intrahepatic Cholestasis; Hepatobiliary Cancer
MeSH Terms: conditions — Cholestasis, Intrahepatic; Cholestasis, progressive familial intrahepatic 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Genotype-phenotype relationship between adult cryptogenic cholestasis and mutations in genes responsible for progressive familial intrahepatic cholestasis

DETAILED DESCRIPTION:
Due to the high number of unsolved cases of adults with cholestatic liver disease, it is crucial to determine the prevalence of PFIC gene mutations and gather information on various clinical presentations that often coexist. This will help identify risk factors related to the disease and its progression, ultimately allowing for personalized treatment options for affected patients.

This multicenter, retrospective observational study will collect data on patients with cholestatic liver diseases (CCLDs) from May 2013 until the study begins. Diagnoses of PFIC/CCLD/HBC will be confirmed through imaging studies, excluding other liver disease causes.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* diagnosis of PFIC/CCLDs/HBCs
* obtaining informed consent

Exclusion Criteria:

* Another documented cause of chronic liver disease capable of justifying the clinical phenotype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data from all patients with PFIC/CCLDs/HBCs will be collected and retrospectively evaluated relating to the centers participating in the study from May 2013 until the start date of the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Mutation classification in PFIC genes in patients with CCLDs | 12 months
  Estimate the percentage of pathological mutations, probably pathological, variants to uncertain significance, probably benign, benign in PFIC genes in subjects with CCLDs

SECONDARY OUTCOMES:
Clinical Outcomes in PFIC Gene Mutation Carriers | 12 months
  Percentage of patients with PFIC gene mutations affected by CCLDs, HBCs, BRIC, LPAC, ICP, DIC, advanced fibrosis, and/or neonatal jaundice
Histological Patterns of Familial Intrahepatic Cholestasis in PFIC Gene Mutation Carriers | 12 months
  Percentages of patients with PFIC genes who have a histological pattern compatible with familial intrahepatic cholestasis.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Vitale, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (2):
- Italy (2):
  - IRCCS - Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - Ospedale Civile Sant'Agostino Estense Baggiovara, Modena, Modena